CLINICAL TRIAL: NCT02906761
Title: Aspirin for Uncontrolled Asthma : a Randomized Controlled Study
Brief Title: Aspirin for Uncontrolled Asthma
Acronym: ASTHMIRINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P130954; 2016-000739-42 (EudraCT Number)
Record Dates: First submitted 2016-09-01; First posted 2016-09-20 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Uncontrolled Asthma
Keywords: asthma, aspirin
MeSH Terms: conditions — Asthma | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): Aspirin 600 mg (2 tablets of 300 mg) twice daily for 6 months
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo (2 tablets) twice daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin 600 mg (2 tablets of 300 mg) twice daily for 6 months
  Other Names: acetylsalicylic acid
  Arms: Aspirin
Drug: Placebo — Placebo (2 tablets) twice daily for 6 months
  Arms: Placebo

SUMMARY:
Asthma is characterized by changes in eicosanoids metabolism, especially high production of bronchoconstrictive cysteinyl leukotrienes (CystLTBs) and leukotriene B4 (LTB4). Recent studies have also demonstrated a relative low production of lipoxin A4, an endogenous lipid mediator resulting from lipo-oxygenase action, distinct from CystLTBs, with anti-inflammatory properties, in bronchial epithelial cells and lung macrophages of severe asthma patients, leading to imbalance between pro-resolving and pro-inflammatory eicosanoids production in airways. Such data suggest that aspirin, that induces lipoxins production, could restore lipoxins deficit in severe asthma. Interest for aspirin is also supported by data obtained in asthma patients with aspirin intolerance (Aspirin induced asthma, AIA) : in this particular group of patients, aspirin treatment significantly improves nasal symptoms, quality of life, asthma and rhinitis scores, and reduces need for hospitalizations, nasal surgery and oral steroids use. Potential effect of aspirin in patients with uncontrolled asthma without aspirin intolerance, who presented changes in arachidonic acid pathway close to those observed in AIA, is not established.

The aim of the study is to assess whether long term aspirin treatment could improve asthma control, compared to placebo, in patients with uncontrolled disease and nasal polyposis, whatever their aspirin tolerance level.

DETAILED DESCRIPTION:
Asthma concerns about 7% of the French adult population. About 10% of them have uncontrolled disease, despite high doses of inhaled steroids combined with long acting beta 2 agonists and adequate management of aggravating factors. They account for considerable asthma morbidity, mortality and costs. New treatments are needed for these patients.

Asthma is characterized by changes in eicosanoids metabolism, especially high production of bronchoconstrictive cysteinyl leukotrienes and LTB4. Recent studies have also demonstrated a relative low production of lipoxin A4, an endogenous lipid mediator resulting from lipo-oxygenase action, distinct from CystLTBs, with anti-inflammatory properties, in bronchial epithelial cells and lung macrophages of severe asthma patients, leading to imbalance between pro-resolving and pro-inflammatory eicosanoids production in airways. Such data suggest that aspirin, that induces lipoxins production, could restore lipoxins deficit in severe asthma, as demonstrated in other models.

Interest for aspirin is also supported by data obtained in asthma patients with aspirin intolerance (Aspirin induced asthma, AIA), who are characterized by a severe difficult-to-treat respiratory disease frequently associated with nasal polyposis, overproduction of leukotrienes and increased expression of leukotriene receptors. In this particular group of patients, aspirin treatment significantly improves nasal symptoms, quality of life, asthma and rhinitis scores, and reduces need for hospitalizations and nasal surgery. A reduction in oral steroids use was observed in most series. In this group of patients, aspirin also induced a decrease in interleukin 4 (IL-4) and Matrix metallopeptidase 9 (MMP-9) levels in sputum in asthma patients thus providing another explanation for anti inflammatory effect of aspirin in asthma. Patients treated with higher doses of aspirin (650 mg BID) had more favorable courses than those treated with lower doses.Aspirin desensitization is considered as a cost-effective therapeutic intervention in patients with moderate-to-severe AIA However, some of these studies, coming mostly from the same team, can be criticized for methodological reasons, low evidence, small series, and weak asthma characterization.

Potential effect of aspirin in patients with uncontrolled asthma without aspirin intolerance, who presented changes in arachidonic acid pathway close to those observed in AIA, is not established. Because similar changes in eicosanoid metabolism are described in nasal polyps mucosa, a pathology frequently associated with asthma, we hypothesize that patients with nasal polyps and asthma could be a specific target for aspirin treatment.

Aspirin is a cheap treatment, compared with biotherapies developed for severe asthma.

Hypothesis The investigators propose to compare the effect aspirin (600 mg twice daily) versus placebo, given during six months, on asthma control in patients with uncontrolled asthma and nasal polyposis, whatever their aspirin level of tolerance, in a randomized, double blind, placebo-controlled trial.

Study objectives Primary objective To assess whether long term aspirin treatment could improve asthma control, compared to placebo, in patients with uncontrolled disease and nasal polyposis, whatever their aspirin tolerance level.

Secondary objectives

To assess the effect of long term aspirin treatment compared to placebo, in patients with uncontrolled disease and nasal polyposis, on the following criteria:

* lung function
* number of exacerbations
* time to the first exacerbation
* oral and inhaled steroid use and doses
* Nasal symptoms
* Nasal sinus symptoms severity
* quality of life
* Lipoxin A4, cysteinyl leukotrienes (cystLT) and LTB4 levels in sputum
* Reactions during oral aspirin challenge
* Gastro-intestinal and other bleedings

Study design This is a multicentric, randomized, placebo-controlled, double-blinded phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 to 75 years old
* Patients receiving inhaled steroids (>1000 µg/d beclomethasone or equivalent) combined with long acting beta agonist at a stable dose for at least 1 month and montelukast for at least 2 weeks.
* Patients receiving Proton Pump Inhibitors for at least 2 weeks
* Uncontrolled asthma defined by an ACQ 6 score≥1.5 at baseline
* Recurrent chronic rhinosinusitis with nasal polyposis diagnosed by nasal endoscopy by an otorhinolaryngologist
* Evidence of reversibility of airway obstruction defined as an increase of FEV1 of 12% or greater and at least 200 ml after Short Acting Beta Agonists (SABA) administration OR after oral corticoid test or an increase of CVF of 12% or greater and at least 200 ml after Short Acting Beta Agonists (SABA) administration or after oral corticoid test OR a variation in FEV1 of more than 200 ml and 12% between 2 follow-up visits OR variation of the Peak Expiratory Flow Rate (PEF) with a delta PEF over the day / average PEF over 2 weeks > 10% OR a positive methacholine bronchial challenge test: decrease in FEV1 by more than 20% for a dose < 1600 µg documented once during medical history
* FEV1>1.5l and 60% of predicted value at inclusion
* Never smoked or non-smoker for at least 6 months, with a smoking history of no more than 10 pack-years
* Written informed consent
* Efficient contraception, other than an intrauterine device (IUD), for women of reproductive age

Exclusion Criteria:

* Evidence of another clinically significant, active pulmonary disorder (bronchiectasis, chronic obstructive pulmonary disease (COPD), …) that could influence asthma control evaluation
* Patient treated regularly with aspirin or NSAID for another pathology
* Hypersensitive response to lansoprazole
* treatment by nelfinavir or other HIV protease inhibitors for which absorption depends on gastric pH (atazanavir...)
* Asthma exacerbation within the 4 weeks prior to inclusion (as defined by an oral corticotherapy for more than 48h or a 2-fold increase of oral corticoid intake )
* Pregnancy or breast feeding
* Recent myocardial infarction within the 6 months prior to inclusion
* immunodeficiency
* Patients receiving bet-blockers
* Contra-indication for aspirin : history of gastro-intestinal or cerebral bleeding, active gastric or duodenal ulcer, major surgery within the 4 weeks prior to inclusion, treatment with methotrexate, probenecid, selective serotonin re-uptake inhibitor, diuretic, angiotensin-converting-enzyme inhibitor, angiotensin receptor inhibitor or anti-platelet drug, ,any hemorrhagic risk according to the investigator, heart, liver or kidney failure, hyperuricemia, phenylketonuria.
* Major surgery planned during the 6 month study period
* under security or legal protection measures
* patient intolerant to lactose or other excipient
* Patient with intra-uterine device
* patient who has not given written consent
* Non affiliation to a social security scheme (beneficiary or assignee)

Secondary exclusion criteria :

-Patients who will require epinephrine injection or transfer to ICU or patients who do not reach the maximum dose of 600mg during aspirin challenge-desensitization will stop the study and not be randomized

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Change in asthma Control Questionnaire (ACQ 6) score between baseline and 6 months | 6 months
  Patients will fill in ACQ6 at each visit (day 0, 1 month, 3 months and 6 months)

SECONDARY OUTCOMES:
Forced expired volume in 1 second (FEV1) variation between baseline and 6 months | 6 months
  A spirometry will be done at each visit (day 0, 1 month, 3 months and 6 months)
number of exacerbations | 6 months
  The number of exacerbations will be assessed at each visit (day 0, 1 month, 3 months and 6 months)
Time to first exacerbation | 6 months
  Time to first exacerbation will be assessed at each visit (day 0, 1 month, 3 months and 6 months)
number of hospitalization | 6 months
  number of hospitalization
oral steroid use | 6 months
  oral steroid use
inhaled steroid doses | 6 months
  inhaled steroid doses
nasal sinus symptoms severity at baseline and 6 months | 6 months
  Patients will fill in Sino-Nasal Outcome Test 16 (SNOT 16) questionnaire at each visit .The SNOT-16 is a quality of life, self-administered questionnaire comprising 16 questions.
  Responses are scored as: 0 = no bother, 1 = mild or minor bother, 2 = moderate bother, 3 = severe bother. Patients are also asked to check to five items which are most important to them personally. Scores range (sum of each question) from 0 (no functional bother) to 48 (maximal functional bother) (day 0, 1 months, 3 months and 6 months)
measure of quality of life: AQLQ | 6 months
  Patients will fill in Asthma Quality of Life Questionnaire (AQLQ) at each visit (day 0, 1 months, 3 months and 6 months). There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). The activity domain contains 5 'patient-specific' questions. This allows patients to select 5 activities in which they are most limited and these activities will be assessed at each follow-up. Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains.
Lipoxin A4 (LXA4) levels in sputum | 6 months
  LXA4 levels at day 0 and 6 months will be measured by ELISA kit
Cyst-LT levels in sputum | 6 months
  Cyst-LT levels at day 0 and 6 months will be measured by ELISA kit
LTB4 levels in sputum | 6 months
  LTB4 levels at day 0 and 6 months will be measured by ELISA kit
Reactions during oral aspirin challenge test | 3 to 4 days
  Occurrence of intolerance symptom : angioedema, bronchospasm, rhinitis, urticaria...
Digestive tolerance during treatment | 6 months
  Medical examination, patient interview
gastro-intestinal bleedings during treatment | 6 months
  Occurence by bleedings during treatment, patient interview

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Service de pneumologie - CHU Besançon, Besançon
  - Service de Pneumologie - Hôpital François Mitterrand - CHU Dijon, Dijon
  - Service de Pneumologie - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Service de pneumologie - Hôpital Calmette - CHRU Lille, Lille
  - Service de Pneumologie - La Croix Rousse, Lyon
  - CIC - Hôpital Bichat, Paris
  - Service de pneumologie - Hôpital Charles Nicolle - CHU Rouen, Rouen
  - Service de pneumologie - Nouvel Hopital Civil - CHU strasbourg, Strasbourg
  - Service de pneumologie - Hôpital Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided